CLINICAL TRIAL: NCT01731873
Title: Non-Interventional Pharmacogenetic Study of Patient / Proxy Controlled Analgesia in Children Undergoing Surgery
Brief Title: Patient Controlled Analgesia Pharmacogenetic Study
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-2268
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Pain
Keywords: postoperative pain; children; pharmacogenetic; opioid adverse effects; respiratory depression; analgesia; genetic polymorphisms; chronic postsurgical pain
MeSH Terms: conditions — Pain; Pain, Postoperative; Respiratory Insufficiency; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A database/ repository will be constructed for future research, analysis, and recruitment. De-identified study participants' genetic information, their responses to pain and pain medications, and side-effects will be included in a study database. Blood specimens will be included in the repository for exploring potentially important SNPs and biomarkers. No patient identifiers will be included in the database, and there will be a confidential (access limited to investigators only) code or link between the database and other information about the participant. Repeat timed blood samples will be collected and analyzed for opioid concentrations and metabolite concentrations (morphine, hydromorphone, fentanyl).
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to identify factors and genes (the nucleic acid material that determines the makeup of the human body) that may be associated with acute and chronic post-surgical pain as well as develop pharmacometric models for response to opioids, like morphine and hydromorphone. While children undergioing different surgeries will be recruited for acute outcomes, children undergoing spine fusion will be followed for 10-12 months for evaluation of psychological and genomic factors affecting chronic post-surgical pain, with a goal of identifying genetic and epigenetic risk models for prediction of acute and chronic post-surgical pain. Although opioids are used every day, some children have bad reactions from their use, like breathing problems, sedation, etc. The investigators want to study factors that may be associated with pain sensitivity, opioid requirements after surgery, their metabolism, efficacy and their side-effects. The investigators expect that the information obtained in this research study will help to develop effective, safer, and tailored treatment options in the future.

DETAILED DESCRIPTION:
Pain management after surgery is not optimal partly due to great interindividual variability in pain perception and coping. This also can lead to persistent pain beyond the healing period and disability. Up to two-thirds of the inter-individual variability result from genetic variations in pain perception as well as response to the pain medicine. The investigators aim to identify genomic (genetic/epigenetic), psychological and drug profiles contributing to this variability. Opioids are the mainstay for treatment of postoperative pain in children. Experience dictates that opioids have narrow therapeutic indices and large inter-patient variability in response. This leads to serious side effects like respiratory depression in up to 50% of children undergoing invasive surgery, which can be fatal. It is evident that there are particular children who are more susceptible to suffering side effects and having inadequate pain relief from opioids.

It is hypothesized that much of the genetic variability can be explained by gene function which is modulated by a) Single Nucleotide Polymorphisms (SNPs) in genes that encode proteins involved in pain perception, opioid transport/metabolism (pharmacokinetics), and opioid receptor signaling (pharmacodynamics); b) epigenetics which modify gene expression without structural changes to the DNA, and c) genes that influence psychological factors.

Identifying genetic and non-genetic predictors for this susceptibility is vital for safe and effective analgesia in children. This is a critical knowledge gap in medical literature that significantly impacts pediatric pain management. The investigators' central hypothesis is that specific genetic polymorphisms in genes involved in pain perception, opioid transport, and opioid receptor signaling pathways contribute significantly to pain sensitivity, opioid side-effects, and analgesic efficacy in children.

The choice and dosing of opioids and pain management approaches have thus far been largely empirical, with a frequent need to switch medications, strategies and alter doses due to inherent differences in individuals. By this study, the investigators hope to develop preemptive approaches and drug targets that can be targeted to individual risk and genomic-psychosocial profiles. The study will help determine the 'right' doses of the 'right' opioids for optimized and safe postoperative analgesia in children. This will be done by first building population pharmacokinetic and pharmacodynamic models for opioid concentration-exposure and then investigating covariates.

Given the unexplored nature of this complex phenomenon, The investigators propose a comprehensive study to evaluate gene, drug, and surgical interactions, in a large sample of 650 children undergoing different surgeries, requiring patient controlled analgesia with opioids.

The investigators' long term goal is to develop more effective, safer, and tailored pediatric opioid analgesia, by contributing to better understanding of the underlying genetic basis for variations in the sensitivity to pain, pain relief, and development of adverse effects from the extended use of postoperative intravenous opioids in children.

The data collected will include acute and long-term pain data, opioid doses, incidence of side-effects of opioids - including respiratory depression, sedation, vomiting, and itching, and blood samples for genetic and pharmacometric analyses. Data analysis will use advanced logistic regression techniques to uncover the association between the SNP variants and the response to specific opioids following various surgeries.

ELIGIBILITY:
Inclusion criteria include:

1. Children up to and including the age of 18 years;
2. Children weighing at least 5kg at time of surgery; and
3. Children scheduled for surgery requiring opioids PCA or PCA by proxy for postoperative pain relief.

Exclusion criteria include:

1. Children with a history of active liver or renal dysfunction (generally indicated by current abnormal lab results);
2. Patients with severe respiratory problems (indicated by an ASA rating > 4, or oxygen/CPAP/BiPAP dependence);
3. Children with recent chronic preoperative pain, especially those requiring opioids or nerve pain medications within the last 6 months prior to surgery;
4. Children who are anticipated to receive ketamine (i.e., injection, infusion, IM) or dexmedetomidine/sufentanil/lidocaine infusions perioperatively;
5. Children with BMI > 35;
6. Children with certain genetic diseases or chromosomal abnormalities known to affect pain perception and/or breathing; and
7. Non-English speaking patients.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (weighing at least 5 kg, and up to and including 18 year olds) undergoing surgery requiring postoperative Patient Controlled Analgesia (PCA) or PCA by Proxy with opioids (P/NCA), shall be eligible for the study, if inclusion/exclusion criteria are met.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 48 hours post-operatively
  Post-surgical pain scores at rest and on mobilization, opioid requirements/48 hours
Chronic post-surgical pain | 6-12 months after surgery
  Pain scores several months after surgery

SECONDARY OUTCOMES:
Opioid pharmacometrics | 24-48 hours postoperatively
  Drug Concentration-Exposure curves
Chronic post-surgical disability | 6-12 months after surgery
  Functional disability scores

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Chidambaran, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with additional internal or external data warehouses/investigators. These include but are not limited to the i2b2-Research Data Warehouse protocol at CCHMC (IRB 2008-0834) for the purpose of linking this data to a de-identified copy of the participant's electronic medical record via an i2b2 database. The resulting de-identified i2b2 database will not be part of this research; but will be used to explore secondary phenotypes in future research studies and documented in the NIH-db-GaP (Database of Genotypes and Phenotypes).

REFERENCES:
- [Background] Sadhasivam S, Boat A, Mahmoud M. Comparison of patient-controlled analgesia with and without dexmedetomidine following spine surgery in children. J Clin Anesth. 2009 Nov;21(7):493-501. doi: 10.1016/j.jclinane.2008.12.017. PMID 20006257
- [Background] Voepel-Lewis T, Marinkovic A, Kostrzewa A, Tait AR, Malviya S. The prevalence of and risk factors for adverse events in children receiving patient-controlled analgesia by proxy or patient-controlled analgesia after surgery. Anesth Analg. 2008 Jul;107(1):70-5. doi: 10.1213/ane.0b013e318172fa9e. PMID 18635469
- [Background] Aubrun F, Monsel S, Langeron O, Coriat P, Riou B. Postoperative titration of intravenous morphine. Eur J Anaesthesiol. 2001 Mar;18(3):159-65. doi: 10.1046/j.0265-0215.2000.00796.x. PMID 11298174
- [Background] Ross JR, Rutter D, Welsh K, Joel SP, Goller K, Wells AU, Du Bois R, Riley J. Clinical response to morphine in cancer patients and genetic variation in candidate genes. Pharmacogenomics J. 2005;5(5):324-36. doi: 10.1038/sj.tpj.6500327. PMID 16103897
- [Background] Ikeda K, Ide S, Han W, Hayashida M, Uhl GR, Sora I. How individual sensitivity to opiates can be predicted by gene analyses. Trends Pharmacol Sci. 2005 Jun;26(6):311-7. doi: 10.1016/j.tips.2005.04.001. PMID 15925706
- [Background] White PF, Kehlet H. Improving postoperative pain management: what are the unresolved issues? Anesthesiology. 2010 Jan;112(1):220-5. doi: 10.1097/ALN.0b013e3181c6316e. No abstract available. PMID 20010418
- [Background] Silverstein JH, Rieders MF, McMullin M, Schulman S, Zahl K. An analysis of the duration of fentanyl and its metabolites in urine and saliva. Anesth Analg. 1993 Mar;76(3):618-21. doi: 10.1213/00000539-199303000-00030. PMID 8452277
- [Background] Feierman DE, Lasker JM. Metabolism of fentanyl, a synthetic opioid analgesic, by human liver microsomes. Role of CYP3A4. Drug Metab Dispos. 1996 Sep;24(9):932-9. PMID 8886601
- [Background] Zanger UM, Turpeinen M, Klein K, Schwab M. Functional pharmacogenetics/genomics of human cytochromes P450 involved in drug biotransformation. Anal Bioanal Chem. 2008 Nov;392(6):1093-108. doi: 10.1007/s00216-008-2291-6. Epub 2008 Aug 10. PMID 18695978
- [Background] Zhang W, Chang YZ, Kan QC, Zhang LR, Li ZS, Lu H, Wang ZY, Chu QJ, Zhang J. CYP3A4*1G genetic polymorphism influences CYP3A activity and response to fentanyl in Chinese gynecologic patients. Eur J Clin Pharmacol. 2010 Jan;66(1):61-6. doi: 10.1007/s00228-009-0726-4. Epub 2009 Sep 26. PMID 19784640
- [Background] D'Arcy Y. One opioid does not fit all. Nurse Pract. 2007 Nov;32(11):7-8. doi: 10.1097/01.NPR.0000298262.47655.14. No abstract available. PMID 18075450
- [Background] Hirota T, Ieiri I, Takane H, Sano H, Kawamoto K, Aono H, Yamasaki A, Takeuchi H, Masada M, Shimizu E, Higuchi S, Otsubo K. Sequence variability and candidate gene analysis in two cancer patients with complex clinical outcomes during morphine therapy. Drug Metab Dispos. 2003 May;31(5):677-80. doi: 10.1124/dmd.31.5.677. PMID 12695358
- [Background] Sadhasivam S, Cohen LL, Szabova A, Varughese A, Kurth CD, Willging P, Wang Y, Nick TG, Gunter J. Real-time assessment of perioperative behaviors and prediction of perioperative outcomes. Anesth Analg. 2009 Mar;108(3):822-6. doi: 10.1213/ane.0b013e318195c115. PMID 19224789
- [Background] Sawyer MB, Innocenti F, Das S, Cheng C, Ramirez J, Pantle-Fisher FH, Wright C, Badner J, Pei D, Boyett JM, Cook E Jr, Ratain MJ. A pharmacogenetic study of uridine diphosphate-glucuronosyltransferase 2B7 in patients receiving morphine. Clin Pharmacol Ther. 2003 Jun;73(6):566-74. doi: 10.1016/S0009-9236(03)00053-5. PMID 12811366
- [Background] Takeda S, Ishii Y, Iwanaga M, Mackenzie PI, Nagata K, Yamazoe Y, Oguri K, Yamada H. Modulation of UDP-glucuronosyltransferase function by cytochrome P450: evidence for the alteration of UGT2B7-catalyzed glucuronidation of morphine by CYP3A4. Mol Pharmacol. 2005 Mar;67(3):665-72. doi: 10.1124/mol.104.007641. Epub 2004 Dec 20. PMID 15611481
- [Background] Beaulieu P, Cyrenne L, Mathews S, Villeneuve E, Vischoff D. Patient-controlled analgesia after spinal fusion for idiopathic scoliosis. Int Orthop. 1996;20(5):295-9. doi: 10.1007/s002640050081. PMID 8930721
- [Background] Duguay Y, Baar C, Skorpen F, Guillemette C. A novel functional polymorphism in the uridine diphosphate-glucuronosyltransferase 2B7 promoter with significant impact on promoter activity. Clin Pharmacol Ther. 2004 Mar;75(3):223-33. doi: 10.1016/j.clpt.2003.10.006. PMID 15001974
- [Background] Benetton SA, Borges VM, Chang TK, McErlane KM. Role of individual human cytochrome P450 enzymes in the in vitro metabolism of hydromorphone. Xenobiotica. 2004 Apr;34(4):335-44. doi: 10.1080/00498250310001657559. PMID 15268978
- [Background] Hanna MH, Elliott KM, Fung M. Randomized, double-blind study of the analgesic efficacy of morphine-6-glucuronide versus morphine sulfate for postoperative pain in major surgery. Anesthesiology. 2005 Apr;102(4):815-21. doi: 10.1097/00000542-200504000-00018. PMID 15791112
- [Background] Smith HS. Opioid metabolism. Mayo Clin Proc. 2009 Jul;84(7):613-24. doi: 10.1016/S0025-6196(11)60750-7. PMID 19567715
- [Background] Shimada T, Yamazaki H, Mimura M, Inui Y, Guengerich FP. Interindividual variations in human liver cytochrome P-450 enzymes involved in the oxidation of drugs, carcinogens and toxic chemicals: studies with liver microsomes of 30 Japanese and 30 Caucasians. J Pharmacol Exp Ther. 1994 Jul;270(1):414-23. PMID 8035341
- [Background] Dahan A, Aarts L, Smith TW. Incidence, Reversal, and Prevention of Opioid-induced Respiratory Depression. Anesthesiology. 2010 Jan;112(1):226-38. doi: 10.1097/ALN.0b013e3181c38c25. PMID 20010421
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] von Baeyer CL, Spagrud LJ, McCormick JC, Choo E, Neville K, Connelly MA. Three new datasets supporting use of the Numerical Rating Scale (NRS-11) for children's self-reports of pain intensity. Pain. 2009 Jun;143(3):223-227. doi: 10.1016/j.pain.2009.03.002. Epub 2009 Apr 8. PMID 19359097
- [Background] Duedahl TH, Hansen EH. A qualitative systematic review of morphine treatment in children with postoperative pain. Paediatr Anaesth. 2007 Aug;17(8):756-74. doi: 10.1111/j.1460-9592.2007.02213.x. PMID 17596221
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Ramsay MA. Anesthesia and pain management at Baylor University Medical Center. Proc (Bayl Univ Med Cent). 2000 Apr;13(2):151-65. doi: 10.1080/08998280.2000.11927660. No abstract available. PMID 16389370
- [Background] Paqueron X, Lumbroso A, Mergoni P, Aubrun F, Langeron O, Coriat P, Riou B. Is morphine-induced sedation synonymous with analgesia during intravenous morphine titration? Br J Anaesth. 2002 Nov;89(5):697-701. PMID 12393765
- [Background] Gramke HF, de Rijke JM, van Kleef M, Raps F, Kessels AG, Peters ML, Sommer M, Marcus MA. The prevalence of postoperative pain in a cross-sectional group of patients after day-case surgery in a university hospital. Clin J Pain. 2007 Jul-Aug;23(6):543-8. doi: 10.1097/AJP.0b013e318074c970. PMID 17575496
- [Background] Sommer M, de Rijke JM, van Kleef M, Kessels AG, Peters ML, Geurts JW, Gramke HF, Marcus MA. The prevalence of postoperative pain in a sample of 1490 surgical inpatients. Eur J Anaesthesiol. 2008 Apr;25(4):267-74. doi: 10.1017/S0265021507003031. Epub 2007 Dec 6. PMID 18053314
- [Background] Fletcher D, Fermanian C, Mardaye A, Aegerter P; Pain and regional anesthesia committee of the French Anesthesia and Intensive Care Society (SFAR). A patient-based national survey on postoperative pain management in France reveals significant achievements and persistent challenges. Pain. 2008 Jul 15;137(2):441-451. doi: 10.1016/j.pain.2008.02.026. Epub 2008 Apr 15. PMID 18417292
- [Background] Brennan F, Carr DB, Cousins M. Pain management: a fundamental human right. Anesth Analg. 2007 Jul;105(1):205-21. doi: 10.1213/01.ane.0000268145.52345.55. PMID 17578977
- [Background] Joshi GP, Kehlet H, Rawal N; PROSPECT Working Group. Evidence-based guidelines for postoperative pain management. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):173. doi: 10.1016/j.rapm.2006.11.002. No abstract available. PMID 17350537
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Chen E, Zeltzer LK, Craske MG, Katz ER. Alteration of memory in the reduction of children's distress during repeated aversive medical procedures. J Consult Clin Psychol. 1999 Aug;67(4):481-90. doi: 10.1037//0022-006x.67.4.481. PMID 10450618
- [Background] D'Arcy Y. Eyeing capnography to improve PCA safety. Nursing. 2007 Sep;37(9):18-9. doi: 10.1097/01.NURSE.0000287701.56255.80. No abstract available. PMID 17728629
- [Background] Maddox RR, Williams CK, Fields M. Respiratory monitoring in patient-controlled analgesia. Am J Health Syst Pharm. 2004 Dec 15;61(24):2628, 2635. doi: 10.1093/ajhp/61.24.2628. No abstract available. PMID 15646697
- [Background] Whitlock MC. Combining probability from independent tests: the weighted Z-method is superior to Fisher's approach. J Evol Biol. 2005 Sep;18(5):1368-73. doi: 10.1111/j.1420-9101.2005.00917.x. PMID 16135132
- [Background] Moore JH, Williams SM. New strategies for identifying gene-gene interactions in hypertension. Ann Med. 2002;34(2):88-95. doi: 10.1080/07853890252953473. PMID 12108579
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Moons KG, Donders AR, Steyerberg EW, Harrell FE. Penalized maximum likelihood estimation to directly adjust diagnostic and prognostic prediction models for overoptimism: a clinical example. J Clin Epidemiol. 2004 Dec;57(12):1262-70. doi: 10.1016/j.jclinepi.2004.01.020. PMID 15617952
- [Background] Nelson KL, Yaster M, Kost-Byerly S, Monitto CL. A national survey of American Pediatric Anesthesiologists: patient-controlled analgesia and other intravenous opioid therapies in pediatric acute pain management. Anesth Analg. 2010 Mar 1;110(3):754-60. doi: 10.1213/ANE.0b013e3181ca749c. PMID 20185654
- [Background] Benhamou D, Viel E, Berti M, Brodner G, De Andres J, Draisci G, Moreno-Azcoita M, Neugebauer EA, Schwenk W, Torres LM. [PATHOS study on postoperative pain management in Europe: French data]. Ann Fr Anesth Reanim. 2008 Sep;27(9):664-78. doi: 10.1016/j.annfar.2008.07.092. Epub 2008 Sep 6. French. PMID 18774676
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Werner MU, Mjobo HN, Nielsen PR, Rudin A. Prediction of postoperative pain: a systematic review of predictive experimental pain studies. Anesthesiology. 2010 Jun;112(6):1494-502. doi: 10.1097/ALN.0b013e3181dcd5a0. PMID 20460988
- [Background] Raja SN, Jensen TS. Predicting postoperative pain based on preoperative pain perception: are we doing better than the weatherman? Anesthesiology. 2010 Jun;112(6):1311-2. doi: 10.1097/ALN.0b013e3181dcd5cc. No abstract available. PMID 20502114
- [Background] Kim H, Ramsay E, Lee H, Wahl S, Dionne RA. Genome-wide association study of acute post-surgical pain in humans. Pharmacogenomics. 2009 Feb;10(2):171-9. doi: 10.2217/14622416.10.2.171. PMID 19207018
- [Background] Skorpen F, Laugsand EA, Klepstad P, Kaasa S. Variable response to opioid treatment: any genetic predictors within sight? Palliat Med. 2008 Jun;22(4):310-27. doi: 10.1177/0269216308089302. PMID 18541635
- [Background] Reyes-Gibby CC, Shete S, Rakvag T, Bhat SV, Skorpen F, Bruera E, Kaasa S, Klepstad P. Exploring joint effects of genes and the clinical efficacy of morphine for cancer pain: OPRM1 and COMT gene. Pain. 2007 Jul;130(1-2):25-30. doi: 10.1016/j.pain.2006.10.023. Epub 2006 Dec 6. PMID 17156920
- [Background] Campa D, Gioia A, Tomei A, Poli P, Barale R. Association of ABCB1/MDR1 and OPRM1 gene polymorphisms with morphine pain relief. Clin Pharmacol Ther. 2008 Apr;83(4):559-66. doi: 10.1038/sj.clpt.6100385. Epub 2007 Sep 26. PMID 17898703
- [Background] Hamburg MA, Collins FS. The path to personalized medicine. N Engl J Med. 2010 Jul 22;363(4):301-4. doi: 10.1056/NEJMp1006304. Epub 2010 Jun 15. No abstract available. PMID 20551152
- [Background] Verghese ST, Hannallah RS. Postoperative pain management in children. Anesthesiol Clin North Am. 2005 Mar;23(1):163-84. doi: 10.1016/j.atc.2004.11.008. PMID 15763417
- [Background] Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Characteristics and prediction of early pain after laparoscopic cholecystectomy. Pain. 2001 Feb 15;90(3):261-269. doi: 10.1016/S0304-3959(00)00406-1. PMID 11207398
- [Background] Keogh E, Herdenfeldt M. Gender, coping and the perception of pain. Pain. 2002 Jun;97(3):195-201. doi: 10.1016/S0304-3959(01)00427-4. PMID 12044616
- [Background] Soetanto AL, Chung JW, Wong TK. Are there gender differences in pain perception? J Neurosci Nurs. 2006 Jun;38(3):172-6. doi: 10.1097/01376517-200606000-00006. PMID 16817669
- [Background] Vargas-Alarcon G, Fragoso JM, Cruz-Robles D, Vargas A, Vargas A, Lao-Villadoniga JI, Garcia-Fructuoso F, Ramos-Kuri M, Hernandez F, Springall R, Bojalil R, Vallejo M, Martinez-Lavin M. Catechol-O-methyltransferase gene haplotypes in Mexican and Spanish patients with fibromyalgia. Arthritis Res Ther. 2007;9(5):R110. doi: 10.1186/ar2316. PMID 17961261
- [Background] Tan EC, Lim Y, Teo YY, Goh R, Law HY, Sia AT. Ethnic differences in pain perception and patient-controlled analgesia usage for postoperative pain. J Pain. 2008 Sep;9(9):849-55. doi: 10.1016/j.jpain.2008.04.004. Epub 2008 Jun 12. PMID 18550441
- [Background] Rahim-Williams FB, Riley JL 3rd, Herrera D, Campbell CM, Hastie BA, Fillingim RB. Ethnic identity predicts experimental pain sensitivity in African Americans and Hispanics. Pain. 2007 May;129(1-2):177-84. doi: 10.1016/j.pain.2006.12.016. Epub 2007 Feb 12. PMID 17296267
- [Background] Kain ZN, Sevarino FB, Rinder C, Pincus S, Alexander GM, Ivy M, Heninger G. Preoperative anxiolysis and postoperative recovery in women undergoing abdominal hysterectomy. Anesthesiology. 2001 Mar;94(3):415-22. doi: 10.1097/00000542-200103000-00009. PMID 11374599
- [Background] Granot M, Ferber SG. The roles of pain catastrophizing and anxiety in the prediction of postoperative pain intensity: a prospective study. Clin J Pain. 2005 Sep-Oct;21(5):439-45. doi: 10.1097/01.ajp.0000135236.12705.2d. PMID 16093750
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Woodhouse A, Ward EM, Mather LE. Intra-subject variability in post-operative patient-controlled analgesia (PCA): is the patient equally satisfied with morphine, pethidine and fentanyl? Pain. 1999 Apr;80(3):545-553. doi: 10.1016/S0304-3959(98)00247-4. PMID 10342416
- [Background] Grass JA. Patient-controlled analgesia. Anesth Analg. 2005 Nov;101(5 Suppl):S44-S61. doi: 10.1213/01.ANE.0000177102.11682.20. PMID 16334492
- [Background] Anderson BJ, Palmer GM. Recent developments in the pharmacological management of pain in children. Curr Opin Anaesthesiol. 2006 Jun;19(3):285-92. doi: 10.1097/01.aco.0000192802.33291.6f. PMID 16735812
- [Background] Sinatra RS, Lodge K, Sibert K, Chung KS, Chung JH, Parker A Jr, Harrison DM. A comparison of morphine, meperidine, and oxymorphone as utilized in patient-controlled analgesia following cesarean delivery. Anesthesiology. 1989 Apr;70(4):585-90. doi: 10.1097/00000542-198904000-00005. PMID 2467588
- [Background] Rakvag TT, Klepstad P, Baar C, Kvam TM, Dale O, Kaasa S, Krokan HE, Skorpen F. The Val158Met polymorphism of the human catechol-O-methyltransferase (COMT) gene may influence morphine requirements in cancer pain patients. Pain. 2005 Jul;116(1-2):73-8. doi: 10.1016/j.pain.2005.03.032. PMID 15927391
- [Background] Nackley AG, Tan KS, Fecho K, Flood P, Diatchenko L, Maixner W. Catechol-O-methyltransferase inhibition increases pain sensitivity through activation of both beta2- and beta3-adrenergic receptors. Pain. 2007 Apr;128(3):199-208. doi: 10.1016/j.pain.2006.09.022. Epub 2006 Nov 7. PMID 17084978
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Background] Coulbault L, Beaussier M, Verstuyft C, Weickmans H, Dubert L, Tregouet D, Descot C, Parc Y, Lienhart A, Jaillon P, Becquemont L. Environmental and genetic factors associated with morphine response in the postoperative period. Clin Pharmacol Ther. 2006 Apr;79(4):316-24. doi: 10.1016/j.clpt.2006.01.007. PMID 16580900
- [Background] Coller JK, Barratt DT, Dahlen K, Loennechen MH, Somogyi AA. ABCB1 genetic variability and methadone dosage requirements in opioid-dependent individuals. Clin Pharmacol Ther. 2006 Dec;80(6):682-90. doi: 10.1016/j.clpt.2006.09.011. PMID 17178268
- [Background] Coffman BL, Rios GR, King CD, Tephly TR. Human UGT2B7 catalyzes morphine glucuronidation. Drug Metab Dispos. 1997 Jan;25(1):1-4. PMID 9010622
- [Background] Darbari DS, van Schaik RH, Capparelli EV, Rana S, McCarter R, van den Anker J. UGT2B7 promoter variant -840G>A contributes to the variability in hepatic clearance of morphine in patients with sickle cell disease. Am J Hematol. 2008 Mar;83(3):200-2. doi: 10.1002/ajh.21051. PMID 17724700
- [Background] Zubieta JK, Heitzeg MM, Smith YR, Bueller JA, Xu K, Xu Y, Koeppe RA, Stohler CS, Goldman D. COMT val158met genotype affects mu-opioid neurotransmitter responses to a pain stressor. Science. 2003 Feb 21;299(5610):1240-3. doi: 10.1126/science.1078546. PMID 12595695
- [Background] Hodges LM, Markova SM, Chinn LW, Gow JM, Kroetz DL, Klein TE, Altman RB. Very important pharmacogene summary: ABCB1 (MDR1, P-glycoprotein). Pharmacogenet Genomics. 2011 Mar;21(3):152-61. doi: 10.1097/FPC.0b013e3283385a1c. No abstract available. PMID 20216335
- [Background] Park HJ, Shinn HK, Ryu SH, Lee HS, Park CS, Kang JH. Genetic polymorphisms in the ABCB1 gene and the effects of fentanyl in Koreans. Clin Pharmacol Ther. 2007 Apr;81(4):539-46. doi: 10.1038/sj.clpt.6100046. Epub 2006 Dec 27. PMID 17192767
- [Background] Ameyaw MM, Regateiro F, Li T, Liu X, Tariq M, Mobarek A, Thornton N, Folayan GO, Githang'a J, Indalo A, Ofori-Adjei D, Price-Evans DA, McLeod HL. MDR1 pharmacogenetics: frequency of the C3435T mutation in exon 26 is significantly influenced by ethnicity. Pharmacogenetics. 2001 Apr;11(3):217-21. doi: 10.1097/00008571-200104000-00005. PMID 11337937
- [Background] Kim RB, Leake BF, Choo EF, Dresser GK, Kubba SV, Schwarz UI, Taylor A, Xie HG, McKinsey J, Zhou S, Lan LB, Schuetz JD, Schuetz EG, Wilkinson GR. Identification of functionally variant MDR1 alleles among European Americans and African Americans. Clin Pharmacol Ther. 2001 Aug;70(2):189-99. doi: 10.1067/mcp.2001.117412. PMID 11503014
- [Background] Diatchenko L, Nackley AG, Slade GD, Bhalang K, Belfer I, Max MB, Goldman D, Maixner W. Catechol-O-methyltransferase gene polymorphisms are associated with multiple pain-evoking stimuli. Pain. 2006 Dec 5;125(3):216-224. doi: 10.1016/j.pain.2006.05.024. Epub 2006 Jul 11. PMID 16837133
- [Background] Weinger M. Dangers of postoperative opioids: APSF Workshop and White Paper address prevention of postoperative respiratory complications. APSF Newsletter 21:61-7, 2006
- [Background] Hutchison R. A Comparison of a Fentanyl, morphine and hydromorphone Patient-controlled intravenous delivery for acute postoperative analgesia: A multicenter study of opioid-induced adverse reactions. Hospital Pharmacy 41:659-63, 2006.
- [Background] Labroo RB, Paine MF, Thummel KE, Kharasch ED. Fentanyl metabolism by human hepatic and intestinal cytochrome P450 3A4: implications for interindividual variability in disposition, efficacy, and drug interactions. Drug Metab Dispos. 1997 Sep;25(9):1072-80. PMID 9311623
- [Background] Radovanovic D. The use of transdermal fentanyl in the treatment of cancer pain. Arch Oncol 10:263-66, 2002.
- [Background] Baselt RC. Disposition of Toxic drugs and Chemicals in Man. 430-33, 2002.
- [Background] Zheng M. Isolation, identification and synthesis of hydromorphone metabolites: analysis and antinociceptive activities in comparison to morphine. 1997.
- [Background] Overdyk M. PCA presents serious risks. APSF Newsletter 20, 2005.
- [Background] D'Argenio DZ, Schumitzky A, Wang X. ADAPT 5 User's Guide: Pharmacokinetic/Pharmacodynamic Systems Analysis Software. Los Angeles: Biomedical Simulations Resource, 2009.
- [Background] D'Argenio D. ADAPT 5 User's Guide: Pharmacokinetic/Pharmacodynamic Systems Analysis Software. Los Angeles: Biomedical Simulations Resource, 2009.
- [Background] Park MY, Hastie T. Penalized logistic regression for detecting gene interactions. Biostatistics. 2008 Jan;9(1):30-50. doi: 10.1093/biostatistics/kxm010. Epub 2007 Apr 11. PMID 17429103
- [Background] Van Slyke DA, Walker LS. Mothers' responses to children's pain. Clin J Pain. 2006 May;22(4):387-91. doi: 10.1097/01.ajp.0000205257.80044.01. PMID 16691093
- [Derived] Chidambaran V, Zhang X, Pilipenko V, Chen X, Wronowski B, Geisler K, Martin LJ, Barski A, Weirauch MT, Ji H. Methylation quantitative trait locus analysis of chronic postsurgical pain uncovers epigenetic mediators of genetic risk. Epigenomics. 2021 Apr;13(8):613-630. doi: 10.2217/epi-2020-0424. Epub 2021 Apr 6. PMID 33820434
- [Derived] Chidambaran V, Ding L, Moore DL, Spruance K, Cudilo EM, Pilipenko V, Hossain M, Sturm P, Kashikar-Zuck S, Martin LJ, Sadhasivam S. Predicting the pain continuum after adolescent idiopathic scoliosis surgery: A prospective cohort study. Eur J Pain. 2017 Aug;21(7):1252-1265. doi: 10.1002/ejp.1025. Epub 2017 Mar 27. PMID 28346762